CLINICAL TRIAL: NCT06723457
Title: A Phase II Study of Combination Epcoritamab-Lenalidomide in Patients With Refractory/Relapsed Immunodeficiency-Related Large B-Cell Lymphoma
Brief Title: Epcoritamab and Lenalidomide in Treating Patients With Refractory or Relapsed Immunodeficiency-Related Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 24H07; NCI-2024-09812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00222751; NU 24H07 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Polymorphic Post-Transplant Lymphoproliferative Disorder; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Specimen Handling; Lenalidomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (epcoritamab, lenalidomide) (Experimental): Patients receive epcoritamab SC weekly during cycle 1 and on days 1, 8, 15, and 22 of cycles 2-3, and day 1 of cycles 4-12. Patients also receive lenalidomide PO on days 1-21 of each cycle. Cycles repeat every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT and collection of blood samples throughout the study and may undergo MRI during screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Epcoritamab; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well the combination of epcoritamab and lenalidomide work in treating patients with immunodeficiency-related large B-cell lymphoma that does not respond to treatment (refractory) or that has come back after a period of improvement (relapsed). Epcoritamab is an immunotherapy that engages T-cells in the immune system to help redirect their killing effects against lymphoma cells. Lenalidomide can modulate the immune system to enhance killing effects of lymphoma by the immune system as well. Giving patients a combination of epcoritamab and lenalidomide may work better in treating refractory or relapsed immunodeficiency-related large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the six-month best response of complete response (CR) rate for the combination of epcoritamab-lenalidomide in chemotherapy ineligible patients with primary refractory or relapsed immunodeficiency-related large B-cell lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate (ORR), partial response (PR) and CR rates at 3 (cycle [C] 4 day [D]1), 6 (C7D1), 12 (30 days post C12), 18 and 24 months for patients on combination epcoritamab-lenalidomide.

II. To assess duration of response (DoR) at 6 (C7D1),12 (30 days post D12), 18 and 24 months for patients on combination epcoritamab-lenalidomide.

III. To assess progression free survival (PFS) with 12,18 and 24 months of follow-up for patients on combination epcoritamab-lenalidomide.

IV. To assess overall survival (OS) with 12, 8 and 24 months of follow-up for patients on combination epcoritamab-lenalidomide.

V. To assess the safety and toxicity of combination epcoritamab-lenalidomide.

EXPLORATORY OBJECTIVES:

I. To assess changes in immune-cell subsets with utilization of epcoritamab-lenalidomide.

II. To evaluate T cell polyfunctionality with the administration of combination epcoritamab-lenalidomide over time.

III. To gain more insights into the phenotype and functional state of different circulating immune cell subsets.

IV. To measure disease-specific symptoms and/or treatment-related concerns in patients treated with combination therapy using Functional Assessment of Cancer Therapy - Lymphoma (FACTLym) European Organization for Research and Treatment of Cancer (EORTC) and Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaires.

OUTLINE:

Patients will receive epcoritamab subcutaneously (SC) weekly during cycle 1 and on days 1, 8, 15, and 22 of cycles 2-3, and day 1 of cycles 4-12. Patients will also receive lenalidomide orally (PO) on days 1-21 of each cycle. Cycles repeat every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients will undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the study and may undergo magnetic resonance imaging (MRI) during screening.

After completion of study treatment, patients will be followed up at 30 days, then at 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of immunodeficiency-related large B-cell lymphoma as defined by the 5th Edition of the World Health Organization (WHO) Classification of Hematolymphoid Tumors 2022 in addition to any of the following:

  * Lymphomas arising in immune deficiency which encompass monomorphic post-transplant lymphoproliferative disorder (PTLD) OR
  * Polymorphic B-cell lymphoproliferative disorder arising in the setting of immunodeficiency and/or immune dysregulation as seen in 1 or more of the following settings:
  * Underlying autoimmune disease
  * Iatrogenic or therapy-related immunosuppression
  * Conditions arising from inborn errors of immunity
  * Immune senescence as seen in patients aged ≥80 years or those ≥ 65 years with CD4 count < 500 cells/mm^3
  * Epstein-Barr virus (EBV) infection as demonstrated by EBV positivity in the tumor cells
* Patients must have measurable disease (≥ 1 measurable nodal lesion [long axis > 1.5 cm] or ≥ 1 measurable extra-nodal lesion [long axis > 1.0 cm] on CT scan or MRI) per Lugano criteria

  * Note; Patients with hepatomegaly /organomegaly deemed to be related to disease will also be eligible if not meeting strict Lugano criteria
* Patients must meet one disease status as follows AND deemed ineligible for chimeric antigen receptor T-cell (CAR-T):

  * Primary refractoriness defined as a partial response or less on interim PET-CT during therapy with frontline chemo-immunotherapy (containing anti-CD20 monoclonal antibody)
  * Primary refractoriness defined as a partial response or less on interim PET-CT during therapy with rituximab (or any other anti-CD20 monoclonal antibody) monotherapy AND deemed ineligible for escalation to chemotherapy
  * Relapse after achieving a complete response with ≥ 1 prior systemic therapy (including CART)
* Patients must be aged ≥ 18 years
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) ≥ 1000/mcL (the use of growth factor support to attain goal ANC allowed, but not the last 14 days prior to screening laboratory test)
* Platelets (PLT) ≥ 50,000/mcL (transfusions allowed ≥ 7 days prior)
* Total bilirubin ≤ 1.5 Institutional upper limit of normal (ULN) unless attributed to Gilbert's ≤ 3 Institutional ULN if attributed to disease or Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional ULN (> 3 and ≤ 5 x institutional upper limit of normal (ULN) if deemed related to disease)
* Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73 m2

  * Estimated (e)GFR is calculated by the abbreviated Modification of Diet in Renal Disease (MDRD)
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of lenalidomide on the developing human fetus are known. For this reason and because lenalidomide as well as other therapeutic agents used in this trial are known to be teratogenic, females of child-bearing potential (FOCBP) must agree to use adequate contraception. Female subjects of reproductive potential must either completely abstain from heterosexual sexual contact or must use 2 effective methods of contraception (at least 1 highly effective method and one effective method) at the same time

  * The 2 effective contraceptive methods must be started at least 30 days before lenalidomide therapy, during therapy (including dose interruptions), and for at least 12 months following discontinuation of therapy
  * Should a female patient become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
  * Females should also refrain from egg donation from the time of informed consent, during the study and for 12 months after the last dose of study drug
  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
  * If male, and subject is sexually active with female partner(s) of childbearing potential, he must agree, from 30 days prior to randomization through 12 months after the last dose of study drug, to practice the protocol-specified contraception
  * Male who is not considering fathering a child or donating sperm during the study or for 12 months after the last dose of study drug
  * FOCBP must have a negative pregnancy test prior to registration on study
* Patients must have no known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

  * (If a patient has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection, the patient must have a negative molecular (e.g., polymerase chain reaction [PCR]) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection)
  * Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations.
  * Patients who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen after they meet the following SARS-CoV-2 infection viral clearance criteria:

    * No signs/symptoms suggestive of active SARS-CoV-2 infection
    * Negative molecular (e.g., PCR) result or 2 negative antigen test results at least 24 hours apart)

Exclusion Criteria:

* Patients who have received any prior therapy with a bispecific T-cell engager targeting CD3 and CD20
* Patients who have received chemotherapy and/or other antineoplastic agents (except CD20- targeting monoclonal antibodies, steroids and/or radiation) within 1 week or 5 half-lives (whichever is shorter) prior to registration
* Patients who have undergone autologous stem cell transplant (ASCT) within 100 days of registration
* Patients who have undergone CAR-T therapy with refractoriness or relapse within 30 days of registration
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to epcoritamab and/or lenalidomide
* Patients with human immunodeficiency virus (HIV) with detectable viral load and CD4 count ≤350 cells/mm3 & not on treatment for more than 1 year
* Patients with evidence of active disease in the central nervous system (CNS) defined as either the presence of active lesions on MRI or cerebrospinal fluid (CSF) studies obtained within 4 weeks prior to registration or progressive neurological decline, attributable to CNS disease
* Patients who have a seizure disorder that is not controlled (requiring anti-epileptic therapy AND with seizure within 12 months of registration)
* Patients who have had major surgery within 4 weeks prior to registration
* Patients who have clinically significant cardiac disease include the following:

  * Myocardial infarction or stroke within 6 months prior to enrollment,
  * OR the following conditions within 6 months prior to enrollment: unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV), uncontrolled cardiac arrhythmia, and uncontrolled hypertension),
  * OR Other clinically significant electrocardiogram (ECG) abnormalities within 6 months prior to enrollment unless deemed stable and appropriately treated
  * OR Left ventricular ejection fraction < 45% for Echocardiogram
* Patients who are unable to swallow, retain and absorb oral tablet/gel/capsules
* Patients who have received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention.

  * Note: Administration of killed vaccines is allowed
* Female patients who are pregnant or nursing.

  * Note: Females should refrain from breast feeding from the time of informed consent, during the study and for 12 months after the last dose of study treatment
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring IV antimicrobial treatment
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-02-18 (Estimated); Study Completion 2029-02-18 (Estimated)

PRIMARY OUTCOMES:
Best response of complete response (CR) rate | At 6 months
  The combination of epcoritamab-lenalidomide in chemotherapy ineligible patients with primary refractory or relapsed immunodeficiency-related large B-cell lymphoma, indicated by the number of patients with CR as best response (using the Lugano Criteria) divided by the total number of patients who have received 1 dose of combination therapy and have had response assessment by radiographic imaging by 6 months from start of therapy. The six-month best response of CR rate will be estimated by the number of patients with complete response divided by the total number of patients who have received 1 dose of combination therapy and have had response assessment by radiographic imaging by 6 months from start of therapy. This estimation will be compared with the historical control 35% by Exact Test of one proportion. At the same time, the Blyth-Still-Casella exact binomial 95% confidence interval of this CR rate will be calculated with adjustment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the initiation of trial therapy until: the response has been confirmed, the subject experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation. This will be assessed at 3, 6, 12, 18, and 24 months.
  The ORR will be estimated by calculating the proportion of treated subjects who experience an objective response (confirmed CR or confirmed partial response [PR] per Lugano Criteria) among all evaluable patients. ORR data will be collected from the initiation of trial therapy (cycle [C] 1 day [D] 1) until: the response has been confirmed, the subject experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first). The ORR, PR and CR rates for patients on combination epcoritamab-lenalidomide, as well as their corresponding Blyth-Still-Casella exact binomial 95% confidence intervals, will be estimated for each time point at 3, 6, 12, 18 and 24 months.
Duration of response (DOR) | The elapses between the day of first documented response to trial therapy (CR or PR, whichever is recorded firstly) and subsequent disease progression, assessed at 6, 12, 18, and 24 months
  The DOR for combination epcoritamab-lenalidomide is defined as the elapses between the day of first documented response to trial therapy (CR or PR, whichever is recorded firstly) and subsequent disease progression (taking as reference for progressive disease the smallest tumor measurements recorded on study per Lugano Criteria), with possible censored at 6, 12, 18, or 24 months for different analysis. By the setting of multiple check and censor time points, the data will be released from cancer center as early as 6 months, which is a routine setting for cellular therapies For DOR analysis, response is defined as CR or PR per the 2014 Lugano Criteria; and disease progression is defined as progressive disease (PD) per the 2014 Lugano Criteria. The median of DOR censored at 6, 12, 18 and 24 months for patients on combination epcoritamab-lenalidomide will be estimated with 95% confidence interval. In addition, the DoRs at different time points will be descrived by Kaplan-Meier curve.
Progression-free survival (PFS) | From initiation of trial therapy to PD per the 2014 Lugano Criteria, other documented clinical or radiographical progression per physician judgement, or death due to disease, assessed at 12, 18, and 24 months
  PFS data will be collected from initiation of trial therapy (C1D1) until the subject suffers disease progression, initiates subsequent anti-cancer therapy due to disease progression on study regimen, completes study participation, or experiences death from any cause (whichever is sooner). If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the PFS will be censored at 12, 18 or 24 months during follow-up. The median of PFS with 12, 18, and 24 months of follow-up for patients on combination epcoritamab-lenalidomide, and corresponding 95% confidence interval, will be estimated. And the Kaplan-Meier curve will be employed again to visualize PFS.
Overall survival (OS) | The time that elapses between initiation of trial therapy and the date of death from any cause for all evaluable patients, assessed at 12, 18, or 24 months.
  OS data will be collected from initiation of trial therapy (C1D1) until the patient completes study follow up participation, experiences death from any cause or is documented as lost to follow up per institutional standard (whichever is sooner). If death from any cause is not observed prior to completing study participation, the OS will be censored as the time of the last available documentation of survival status. The median of OS with 12, 18, and 24 months of follow-up for patients on combination epcoritamab-lenalidomide, and corresponding 95% confidence interval, will be estimated. And the Kaplan-Meier curve will be employed again to visualize OS.
Incidence of adverse events | Up to 24 months
  The toxicity profile of each study drug and combination of study drugs will be assessed. This endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution to one or both, according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States